CLINICAL TRIAL: NCT02751437
Title: Effect of Preterm Arginine INTake on Biological Pathways Affecting Immune Function in Infants Requiring Early Parenteral Nutrition
Brief Title: Preterm Arginine INTake Study
Acronym: PAINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool Women's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LWH1077
Record Dates: First submitted 2016-03-21; First posted 2016-04-26 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Preterm Infant Nutrition and Immune Function
Keywords: preterm; arginine; immune function; nutrition
MeSH Terms: conditions — Premature Birth | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Arginine unsupplemented (No Intervention): These infants identified as having low blood arginine levels will receive standard care.
- Low Arginine supplemented (Experimental): These infants identified as having low arginine levels will receive an additional arginine infusion between days 3 and 10 of life.
  Interventions: Dietary Supplement: Arginine
- Normal Arginine (No Intervention): These infants identified as having normal arginine levels will receive standard care.

INTERVENTIONS:
Dietary Supplement: Arginine
  Arms: Low Arginine supplemented

SUMMARY:
The investigators will explore the effect of current intravenous feeding (parenteral nutrition (PN)) formulations on blood arginine levels and the genes that are involved in body nutrition and fighting infection in premature babies. They will also investigate the effect of supplementing arginine on these genes. The investigators will undertake a single centre exploratory physiological study in 12 very premature infants receiving PN. 4 of these infants will be supplemented with arginine. The investigators will record nutritional intake and routine biochemical testing data (which includes amino acid levels) collected over the first 10 days of life. They will take blood for analysis at prespecified intervals for microarray, ammonia and IGF-1 levels. Microarray findings will allow the investigators to describe the effect of arginine on gene activity in preterm infants.

DETAILED DESCRIPTION:
Title:

Effect of Preterm Arginine INTake on biological pathways affecting immune function in infants requiring early parenteral nutrition (PAINT)

Population: Preterm infants <29 weeks gestation

Number of infants: 12 infants (completing the study) will be recruited over approximately 12 months

Number of sites: One. Infants will be born at Liverpool Women's Hospital (LWH) or transferred to LWH within 48 hours of birth.

Study duration: Informed consent will take place within 72 hours of birth. The first study related blood sample will be taken at this point and will determine arginine status (using blood ammonia and arginine levels) with the last sample taken on postnatal day 10. Other study assessments reflect those routinely performed in preterm infants receiving parenteral nutrition (PN).

Study intervention: All infants will receive standard clinical treatment. The study will involve 4 infants with normal arginine status, and 8 infants with evidence of arginine deficiency. Of these, 4 infants will receive standard PN and the study intervention of an additional arginine infusion of 10mg/kg/hr from day 3 until day 10, the other 8 infants will receive standard PN only.

Primary objective: To determine the alterations in gene expression present in infants <29 weeks gestation (and shown to be arginine deficient on day 3) between day 3 and day 10 in infants receiving additional arginine supplementation. The changes in gene expression will be compared with those seen between day 3 and day 10 in unsupplemented infants, with and without arginine deficiency. The genes of interest are those involved in T-cell function and associated inflammatory pathways.

Secondary objectives:

1. To explore other biological pathways i) known to be involved in the pathogenesis of necrotising enterocolitis ii) involved in arginine metabolism iii) that are related to the insulin-IGF-I axis
2. To assess whether there is an association between high ammonia levels (as a measure of functional arginine deficiency) and T-cell dysfunction and associated inflammatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 23 and 29 completed weeks gestation and admitted to the neonatal unit within 48 hours of birth

Exclusion Criteria:

* Infants who are unlikely to survive the first week after birth.
* Infants with early onset infection (<72 hours)
* Infants known (or suspected to have) a diagnosis of inborn error of metabolism or serious liver dysfunction
* Parents who are unable to give informed consent

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
The pattern of alteration in gene expression between day 3 and day 10 in arginine deficient preterm infants after supplementation with arginine. | Samples on Day 3 and Day 10 of life
  The changes in gene expression will be compared with those seen in unsupplemented infants, with and without arginine deficiency. The genes of interest are those involved in T-cell function and associated inflammatory pathways.

SECONDARY OUTCOMES:
The pattern of alteration in gene expression associated with biological pathways known to be associated with NEC. | Day 3 and Day 10 of life
The pattern of alteration in gene expression associated with biological pathways known to be involved in arginine metabolism | Day 3 and Day 10 of life
The pattern of alteration in gene expression associated with biological pathways that are related to the IGF-1-insulin axis | Day 3 and Day 10 of life
To validate if high ammonia levels (as a measure of functional arginine deficiency) are linked with impaired T-cell function and associated inflammatory pathways | Day 3 of life

CONTACTS AND LOCATIONS:
Overall Officials: Colin Morgan, MBBS BSc MD, Study Director — Neonatal Unit, Liverpool Women's Hospital, Crown St, Liverpool, L8 7SS
Locations (1):
- Liverpool Women's Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available